CLINICAL TRIAL: NCT00699920
Title: A Randomised Study to Compare a Fixed Dose Combination of Artesunate Plus Amiodaquine (Coarsucam) Versus a Fixed Dose Combination of Artemether Plus Lumefantrine (Coartem) in the Treatment of Repeated Uncomplicated Plasmodium Falciparum Malaria Attacks Occurring During the 2 Years of Follow-up, in Children in Uganda.
Brief Title: Cohort Study in Uganda Comparing Artesunate + Amiodaquine (Coarsucam) Versus Artemether + Lumenfantrine (Coartem) in the Treatment of Repeated Uncomplicated Plasmodium Falciparum Malaria Attacks
Acronym: SMART-CURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAMF_L_02661
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

ARMS (2):
- 1 (Experimental): Coarsucam double-layer artesunate/amiodaquine tablets
  Interventions: Drug: Coarsucam
- 2 (Active Comparator): Coartem (artemether/lumefantrine) fixed-dose combination tablets
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: Coarsucam — Oral route, once daily, dose according to bodyweight range Duration of treatment: 3 days
  Arms: 1
Drug: Coartem — Oral route, twice daily, dose according to bodyweight range Duration of treatment: 3 days
  Arms: 2

SUMMARY:
Primary objective is to demonstrate the non-inferiority of PCR (Polymerase Chain Reaction) adjusted adequate clinical and parasitological response at Day 28 of Coarsucam versus Coartem, based on the first malaria attack of each patient.

Secondary objectives:

For the first attack:

To compare the 2 groups of treatment in terms of:

* Day 42 efficacy
* Parasitological and fever clearance
* Clinical and Biological tolerability
* Evolution of gametocyte carriage

For attack 2nd and following:

To compare the 2 groups of treatment in terms of:

* Day 28 and Day 42 clinical and parasitological effectiveness
* Clinical and Biological tolerability
* Proportion of patients without fever at Day 3
* Proportion of patients without parasites at Day 3
* Evolution of gametocyte carriage
* Compliance

During the total follow up of the cohort:

To compare the 2 groups of treatment in terms of:

* Treatment incidence density
* Impact of repeated treatment on clinical and biological tolerability
* Impact on anaemia
* Impact on Hackett score.

ELIGIBILITY:
Inclusion Criteria:

Specific inclusion criteria for initial enrollment:

* Confirmed mono infection with Plasmodium falciparum, with parasite density ≥2000 asexual forms per µl of blood,

Inclusion criteria for each attacks:

* Body weight ≥5 kg
* Able to be treated by oral route
* Fever (axillary temperatur ≥37.5 degrees Celsius) at D0 or history of fever within the previous 24 hours
* Confirmed Plasmodium falciparum infection with positive paratesimia
* Haemoglobin value ≥5.0 g/dl

Exclusion Criteria:

Specific exclusion criteria for initial enrollment:

* Patient participating in another ongoing clinical trial
* Allergy to one of the investigational medicinal products
* History of hepatic and (or) haematological impairment during treatment with amodiaquine
* History of cardiac disease
* Concomitant febrile illness

Exclusion criteria for each attacks:

* Presence of at least one danger sign of malaria: recent history of convulsions (1-2 within 24h), unconsciousness state, lethargy, unable to drink or breast feed, vomiting everything, unable to stand/sit due to weakness
* Severe concomitant disease or known disturbances of electrolyte balance such as hypokalaemia or hypomagnesaemia
* Intake of medication metabolized by cytochrome CYP 2D6 (e.g. metoprolol, flecainide, imipramine, amitriptyline, clomipramine) at the time of inclusion
* Intake of drugs known to inhibit CYP 2A6 (e.g. methoxsalem, pilocarpine, tranylcypromine) and/or 2C8 cytochromes (e.g. trimethoprim, ritonavir, ketoconazole, montelukast, gemfibrozil) at the time of inclusion
* Intake of medication known to prolong the QTc interval, such as class IA and III antiarrythmics, neuroleptics, antidepressant agents, certain antibiotics including drugs in the macrolide class, fluoroquinolones, imidazole and triazole, antifungal agents, certain non-sedative anthistamines (terfenadine, astemizole) and cisapride at the time of inclusion
* Patient having received artesunate + amiodaquine or artemether + lumefantrine at suitable dosage within the previous 2 weeks.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 413 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PCR corrected and uncorrected clinical and parasitological cure rate | At Day 28

SECONDARY OUTCOMES:
Fever and parasitological clearance evaluation by measuring the axillary temperature and monitoring paratesimia | At the first attack
Proportion of afebrile patients and proportion of patients without parasites | At Day 3 (following attacks)
Evolution of baseline symptoms (Clinical efficacy measure) | During the study conduct
Number of residual tablets in blisters (compliance) | At the end of the study treatment
Treatment incidence density: comparison of the number of malaria attacks between the 2 arms | During the 2 years of follow-up
Mean delay between 2 attacks | during the 2 years of follow-up
Incidence and intensity of recorded AE | from the informed consent signed up to the end of the study
Biological tolerability (Hb, Bilirubin, ALAT, Creatinine, Leucocytes, Neutrophils and Platelets count) | During the study conduct
PCR corrected and uncorrected clinical and parasitological cure rate | At Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lemeyre, Study Director — Sanofi
Locations (1):
- Sanofi-aventis administrative office, Kampala, Uganda

REFERENCES:
- [Derived] Yeka A, Lameyre V, Afizi K, Fredrick M, Lukwago R, Kamya MR, Talisuna AO. Efficacy and safety of fixed-dose artesunate-amodiaquine vs. artemether-lumefantrine for repeated treatment of uncomplicated malaria in Ugandan children. PLoS One. 2014 Dec 1;9(12):e113311. doi: 10.1371/journal.pone.0113311. eCollection 2014. PMID 25436614